CLINICAL TRIAL: NCT04429347
Title: Effect of Gabapentin and Tizanidine on Insomnia in Chronic Pain Patients: A Randomized, Double-blind, Placebo-controlled Crossover Trial.
Brief Title: Gabapentin and Tizanidine for Insomnia in Chronic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Nathaniel Schuster, Assistant Profesor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 191167; UL1TR000100 (NIH)
Record Dates: First submitted 2020-05-22; First posted 2020-06-12 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Insomnia Due to Medical Condition; Chronic Pain
Keywords: Insomnia; Chronic Pain; Gabapentin; Tizanidine; Placebo
MeSH Terms: conditions — Chronic Pain; Sleep Initiation and Maintenance Disorders | interventions — Gabapentin; salicylhydroxamic acid; Sugars; tizanidine

STUDY DESIGN:
Intervention Model Description: Randomized, Double-bind, Placebo-controlled, Crossover Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each participant will have an identification number and randomization of drug sequence allocation will be performed a priori using a random number generator by the study pharmacist. The 3 treatments will be identically encapsulated by the study pharmacist. The study pharmacist will place the drug capsules in identical sealed plastic bags labeled "Treatment 1" through "Treatment 3".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Tizanidine 2mg (Experimental): Friday night: 1 capsule Saturday night: 2 capsules Sunday night: Subject chooses 1-2 capsules
  Interventions: Drug: Tizanidine
- Gabapentin 300mg (Experimental): Friday night: 1 capsule Saturday night: 2 capsules Sunday night: Subject chooses 1-2 capsules
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): Friday night: 1 capsule Saturday night: 2 capsules Sunday night: Subject chooses 1-2 capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — Friday night: 1 capsule of 300 mg, Saturday night: 2 capsule of 300 mg (total 600 mg), Sunday night: choice of 1 or 2 capsule of 300 mg (total of 300 or 600 mg)
  Other Names: Neurontin
  Arms: Gabapentin 300mg
Drug: Placebo — Friday night: 1 capsule, Saturday night: 2 capsule, Sunday night: choice of 1 or 2 capsules
  Other Names: Sham; Sugar Pill
  Arms: Placebo
Drug: Tizanidine — Friday night: 1 capsule of 2 mg, Saturday night: 2 capsule of 2 mg (total 4 mg), Sunday night: choice of 1 or 2 capsules of 2 mg (total of 2 or 4 mg)
  Other Names: Zanaflex
  Arms: Tizanidine 2mg

SUMMARY:
This is a double-blind, placebo-controlled, randomized, crossover trial aimed at assessing the effect of gabapentin and tizanidine, two pain medications, on insomnia in chronic pain patients.

DETAILED DESCRIPTION:
Chronic pain and insomnia are highly prevalent conditions affecting 10-25% and 6-10% of the general population, respectively. Importantly, these two conditions frequently co-occur, with 50-80% of chronic pain patients reporting sleep disturbances. Identifying medication that alleviates pain and insomnia simultaneously may help reduce risks associated with polypharmacy, including drug-drug interactions.

In this double-blind, placebo-controlled, randomized, crossover trial, gabapentin and tizanidine, two drugs which are respectively commonly used to treat neuropathic and musculoskeletal pain, will be compared to each other and to placebo in their ability to alleviate insomnia in chronic pain patients.

In each week, patients will receive 3-night (Friday-Sunday) trials each of placebo, gabapentin or tizanidine in a randomized, double-blind order and will monitor their insomnia using the Athens Insomnia Scale (AIS) questionnaire (adapted to fit the time frame of this trial). The primary outcome consists of the difference in mean AIS scores between the 3 treatments at the primary time point, which is Monday of each week (after 3 nights of drug intake).

Patients will also monitor their sleepiness, pain relief and overall improvement as secondary variants using the Stanford Sleepiness Scale (SSS), Visual Analog Scale (VAS), and Patient's Global Impression of Change (PGIC) questionnaires respectively.

Scores on the Monday preceding the first treatment will serve as baseline and the period between treatments (i.e. Monday-Thursday nights) will serve as a 4-day washout period between treatments.

Our hypothesis is that gabapentin and tizanidine will both be more effective than placebo in alleviating insomnia in chronic pain patients but will not be different from one another.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≤ 35
* Any ethnicity
* Must be able to communicate in English
* Must have access to email and be able to respond to REDCap questionnaires in English
* Has a chronic pain condition (≥ 3 months of pain)
* Reports sleep disturbance and scores ≥ 6 on AIS questionnaire
* Ability to provide informed consent

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Has diagnosis of chronic kidney disease
* Has known QT prolongation >500 msec on prior EKG
* Inability to complete daily questionnaires
* Allergy to, or intolerance of, any of tizanidine or gabapentin
* Shift workers
* Anticipated travel across multiple time zones (jetlag) during the duration of the trial
* Circadian misalignment
* Prior syncope experience and/or fear of blood/needles (if a blood draw is required)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Sleep quality | Monday after 3 nights of drug intake
  Comparison of group means for Athens Insomnia Scale scores between the 3 treatment groups placebo, gabapentin and tizanidine.
  Total Athens Insomnia Scale score ranges from 0 to 24. The higher the score, the more severe the insomnia symptoms experienced by the patient.

SECONDARY OUTCOMES:
Pain Intensity | Monday after 3 nights of drug intake
  Comparison of group means for Visual Analog Scale scores between the 3 treatment groups placebo, gabapentin and tizanidine.
  Visual Analog Scale score ranges from 0 to 10. The higher the score, the worse the pain experienced by the patient.
Alertness | Monday after 3 nights of drug intake
  Comparison of group means for Stanford Sleepiness Scale scores between the 3 treatment groups placebo, gabapentin and tizanidine.
  Stanford Sleepiness Scale score ranges from 1 to 7. The higher the score, the more sleepy and less alert the patient.
Overall improvement | Monday after 3 nights of drug intake
  Comparison of group means for Patient Global Impression of Change scores between the 3 treatment groups placebo, gabapentin and tizanidine.
  Patient Global Impression of Change score ranges from 1 to 7. The higher the score, the more improvement reported by the patient.
Categorical assessment of insomnia improvement | Monday after 3 nights of drug intake
  Percentage of patients with a 30% improvement from baseline in individual Athens Insomnia Scale scores for each of the 3 treatments placebo, gabapentin and tizanidine.
  Total Athens Insomnia Scale score ranges from 0 to 24. The higher the scores, the more severe the insomnia symptoms experienced by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Schuster, MD, Principal Investigator — UC San Diego
Locations (1):
- Center for Pain Medicine, UC San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared in a manner TBD based on funding availability and journal requirements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 12 months and ending 3 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be sent to nmschuster@health.ucsd.edu.